CLINICAL TRIAL: NCT00558857
Title: Clinical Feasibility of Using Dynamic Substrate Mapping to Guide Ablation of Ischemic Ventricular Tachycardia
Brief Title: Dynamic Substrate Mapping (DSM) for Ischemic VT
Acronym: DSM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Donna Godejohn, St. Jude Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 065.5
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Ventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSM (Active Comparator): Treatment using DSM to guide ablation
  Interventions: Device: Dynamic Substrate Mapping-guided ablation

INTERVENTIONS:
Device: Dynamic Substrate Mapping-guided ablation — Radiofrequency ablation

SUMMARY:
This is a prospective, non-randomized study to determine the feasibility of using a new technique called Dynamic Substrate Mapping (DSM) to help guide the treatment of ischemic ventricular tachycardia (IVT). We hypothesize that DSM will lead to simpler, more effective ablation of IVT. Results from this study will be used to determine if further clinical investigation is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Have an ICD or CRT-D device
* Had at least 3 documented device therapies to treat VT over last 3 months
* Clinical VT is confirmed or suspected to be of ischemic origin
* Scheduled for VT ablation procedure
* LVEF > or = 20%

Exclusion Criteria:

* Inadequate AAD washout (amiodarone should be maintained at current dose)
* Unstable angina
* Active ischemia
* Cardiac surgery within prior 2 months
* Evidence of infection
* Prosthetic mitral or aortic valve or mitral/aortic valvular heart disease requiring surgical intervention
* History of embolic event
* Myocardial infarction within prior 6 weeks
* Enrolled in another study
* Recurrent sepsis or otherwise not a candidate for catheterization
* Hypercoagulable state or inability to tolerate heparin therapy during procedure
* Has had an atriotomy or ventriculotomy within prior 4 months
* Life expectancy < 6 months
* Class IV NYHA classification

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David Callans, MD, Principal Investigator — University of Pennsylvania; Jason Jacobson, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia